CLINICAL TRIAL: NCT02169076
Title: Cardiac Resynchronization Therapy in Patients With Left Ventricular Assist Devices
Brief Title: Impact of Cardiac Resynchronization Therapy on Right Ventricular Function in Left Ventricular Assist Device Patients
Acronym: CRT-LVAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Approval withdrawn
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14.0338
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
Keywords: Ventricular Assist Device, Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-On (Active Comparator): Cardiac Resynchronization Therapy enabled on ICD/Pacemaker device
  Interventions: Device: Cardiac Resynchronization Therapy
- CRT-Off (Sham Comparator): Cardiac Resynchronization Therapy disabled on ICD/Pacemaker device
  Interventions: Device: Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — The cardiac resynchronization therapy of the ICD/Pacemaker device of the patients enrolled in the study will be programed under a standardized protocol and enabled or disabled in a crossover fashion during the study.

SUMMARY:
Left Ventricular Assist Devices (LVAD) are mechanical heart pumps that are increasingly being implanted in patients with severe heart failure which have failed medical therapy. In patients with LVADs, right ventricular failure, which is not supported by the LVAD pump, is a major problem that affects quality-of-life and survival. Cardiac Resynchronization Therapy (CRT) aims to restore the synchronized contraction of the heart and has proven to be beneficial for improving ejection fraction of both right and left ventricle as well as quality of life in selected heart failure patients. The role of CRT in patients with LVADs is unknown. We hypothesize that CRT can exert a beneficial impact on right ventricular function in LVAD patients and improve their quality-of-life.

The specific questions that this study aims to answer are:

1. What are the effects of CRT on the function of the non-supported right ventricle in patients with an implanted LVAD?
2. Can the effects of CRT on cardiac function positively impact quality-of-life and exercise capacity in LVAD recipients?

In this study patients with a previously implanted CRT device, who later receives an LVAD, will be randomly assigned to have the CRT turned off (CRT-off) or on (CRT-on). The patients will be followed for an 8-week period, and then switched over to the opposite CRT status. The total participation in this study will last for 16 ± 1 weeks, and will involve 3 clinic visits of approximately 3 hour duration (initial visit, 8 week visit, and 16 week final visit), plus 2 quick checks of the pacemaker/defibrillator in-between the visits. Heart function will be assessed with comprehensive echocardiographic studies during the CRT "on" and CRT "off" periods. Quality-of-life and exercise capacity will be assessed with a standardized questionnaire and a 6-Minute Walk Test.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with previously implanted Bi-Ventricular pacemaker / defibrillator, and continuous flow LVAD (Heart Mate II® or HeartWare®)
* The LVAD must be implanted between 8 weeks and 18 months prior to enrollment
* Patients should be at least 3 weeks post discharge from the LVAD implant hospitalization

Exclusion Criteria:

* Severe decompensated right ventricular failure defined as requiring any of the following:

  * Hospitalization for heart failure within last 30 days
  * Need for inotropic infusion for > 48h within the last 14 days
  * Increase of > 100% diuretic dose within last 14 days
* Severe aortic regurgitation documented by echocardiography or cardiac catheterization
* Stage IV or greater kidney disease (GFR < 30 mL/min/1.73 m2)
* Active infection (not including controlled chronic driveline infection on suppressive antibiotic therapy)
* Biventricular pacing < 90 % of time due to uncontrolled arrhythmias
* LVAD malfunction
* Inability to follow study protocol
* Non-functional LV lead (i.e. high capture threshold that cannot be corrected with programming changes)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Right ventricular function | 8 weeks
  The primary cardiac performance endpoint is global longitudinal right ventricular (RV) function assessed by myocardial strain analysis using Speckle Tracking Echocardiography (STE).
  Other traditional echocardiographic RV function indexes will also be evaluated.

SECONDARY OUTCOMES:
Functional capacity | 8 weeks
  Will be assessed by 6-Minute Walk Test

OTHER OUTCOMES:
Quality-of-Life | 8 weeks
  Assessed by standardized self administered Minnesota Living with Heart Failure Questionnaire (MLHFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Gopinathannair, MD, MA, FHRS, Principal Investigator — University of Louisville; Martin A Espinosa Ginic, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States